CLINICAL TRIAL: NCT01773356
Title: Randomized, Controlled, Parallel Trial to Evaluate the Effects of Dihydrocapsiate on Energy Expenditure in Women
Brief Title: Effect of Dihydrocapsiate on Energy Expenditure in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellen Evans (Other)
Collaborators: Kellogg Company (Industry)
Responsible Party: Sponsor-Investigator, Ellen Evans, Dr Ellen Evans, University of Georgia
Organization: University of Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WASABI
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: Obesity; Body Weight; Body Composition; Metabolism; Resting Energy Expenditure
MeSH Terms: conditions — Obesity; Body Weight | interventions — capsiate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo 0 mg/d (Placebo Comparator): 0 mg/d of Dihydrocapsiate will be consumed in ready to ear cereal, cereal bars or crackers
  Interventions: Dietary Supplement: Dihydrocapsiate
- Dihydrocapsiate 9 mg/d (Active Comparator): 9 mg/d of Dihydrocapsiate will be consumed in ready to ear cereal, cereal bars or crackers
  Interventions: Dietary Supplement: Dihydrocapsiate

INTERVENTIONS:
Dietary Supplement: Dihydrocapsiate — Kellogg's ready to eat cereal, cereal bars, and crackers will contain dihyrocapsiate or placebo. Daily consumption of dihydrocapsiate is 9mg/d or 0mg/d.
  Other Names: Natural substances present in sweet chili peppers

SUMMARY:
The objective of this study is to test the effect of dihydrocapsiate on energy expenditure in women.

DETAILED DESCRIPTION:
Capsaicin, a substance found in chili pepper, is known to stimulate thermogenesis. Dihydrocapsiate, a capsinoid, found in the non-pungent CH-19 sweet pepper has similar thermogenic effects without the gastrointestinal side effects. The objective of this project is to test the effect of 12 weeks of daily consumption of 9 mg dihydrocapsiate on resting energy expenditure relative to baseline when compared to a control group consuming products without DCT.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-34.5 kg/m2
* Good general health
* Low to mild physical activity
* Willing to maintain habitual diet and physical activity patterns throughout the study period
* Premenopausal and cycling regularly or using oral contraceptives
* Willing to attend study visits only during the follicular phase or bleed phase of their menstrual cycle
* Understands study procedures and signs forms providing informed consent to participate in the study
* Have spoken and written English literacy

Exclusion Criteria:

* Diabetes mellitus or any conditions that might affect energy metabolism
* Weight change ±2 kg over previous three months
* Known sensitivity or allergy to ingredients of the study products
* Non-breakfast eater
* Recent use of antibiotics
* History of smoking during the six months prior to study
* Recent signs or symptoms of infection, including cold or flu-like symptoms
* Concurrent or recent intervention study participation
* Instability in breathing patterns or energy expenditure measures
* History of drug or alcohol abuse
* Lipid-lowering, anti-hypertensive or anti-inflammatory steroid medication use
* Weight loss medication
* Pregnant or lactating
* Unwilling to be randomized to any experimental group and unable to meet all requirements of the study

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | Change from Baseline at 12 weeks

SECONDARY OUTCOMES:
Thermic effect of feeding | Change from baseline at 12 weeks
Body Composition | Change from baseline at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Evans, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Department of Kinesiology, Athens, Georgia, United States